CLINICAL TRIAL: NCT03337360
Title: The Impact of a Nutritional Supplement (Impryl®) on Male Fertility
Acronym: SUMMER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Goodlife Fertility B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL61414.091.17; NTR6551 (Registry Identifier: Nederlands Trial Register)
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Male Subfertility
Keywords: fertility; male subfertility; foodsupplement; oxidative stress
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised double blind placebo controlled clinical trial/superiority study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impryl (Active Comparator): One tablet daily for 6 months
  Interventions: Dietary Supplement: Impryl
- Placebo (Placebo Comparator): One tablet daily for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Impryl — Food supplement with betaine, cystine, zinc, niacin, folic acid (5MTHF-glucosamine), Vitamin B12 (cobalamin), Vitamin B6, Vitamin B2 (riboflavin)
  Arms: Impryl
Other: Placebo — Inactive ingredients, placebo
  Arms: Placebo

SUMMARY:
Infertility is a worldwide problem and about 10%-15% of all couples will be affected by the inability to have children. In approximately 50% of infertile couples a male factor is involved. Male infertility is of multifactorial origin. In the past decade, the role of oxidative stress on sperm has been researched thoroughly and found to be the problem in 30% to 80% of male infertility cases.

Impryl® is a nutritional supplement mainly consisting of vitamin B, which works on the metabolic system by activating the one carbon cycle and recycling of homocysteine without the use of any direct strong antioxidants.

In this study the investigators want to determine the effectiveness of nutritional supplement Impryl® in men of infertile couples on ongoing pregnancy rate, with or without assisted reproduction technology (ART).

DETAILED DESCRIPTION:
Rationale: Infertility is a worldwide problem and about 10%-15% of all couples will be affected by the inability to have children. In approximately 50% of infertile couples a male factor is involved. In the past decade, the role of oxidative stress on sperm has been researched thoroughly and found to be the problem in 30% to 80% of male infertility cases. Impryl® is a nutritional supplement which works on the metabolic system and regulation of oxidative stress by activating the 1-Carbon cycle and therefore recycling of homocysteine.

Objective: To determine the effectiveness of nutritional supplement Impryl® in men of infertile couples on ongoing pregnancy rate, with or without assisted reproduction technology (ART).

Study design: Multicentre, randomised double blind placebo controlled clinical trial/superiority study.

Study population: All participants in this study are male adults, age 18-50 years, part of a couple that is diagnosed with infertility, regardless the outcome of semen analysis. The couple will either start or is already started with fertility treatment, i.e. expectative management (EM, duration 6 months), intra-uterine insemination (IUI) with or without ovarian stimulation (mild ovarian hyperstimulation (MOH) or ovulation induction (OI)), either in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) treatment.

Intervention: Impryl® or placebo, with identical appearance one tablet each day for a total duration of maximal 6 months. Patients can start directly with study medication and fertility treatment (or to conceive spontaneously).

Main study parameters/endpoints: The primary outcome is the number of ongoing pregnancies confirmed by ultrasound at ≥ 10-12 weeks. Secondary outcomes are change in semen parameters between baseline and 3 months intervention in IUI/IVF/ICSI group, based on (pre-wash) total motile sperm count (TMSC), leading to a change in treatment category Furthermore the occurrence of pregnancy, time to pregnancy, embryo fertilization rate in IVF/ICSI, embryo-utilization rate in IVF/ICSI, number of miscarriages and live birth rate are documented within the study period. The occurrence of adverse events will be reported.

ELIGIBILITY:
Inclusion Criteria:

Couples with failure to conceive for at least 12 months and starting with EM or Couples starting with 1st/ 2nd/3rd cycle of IUI (with/without ovarian stimulation) or Couples starting with 1st/ 2nd/3rd cycle of IVF/ICSI

Furthermore:

* Male with age 18-50 years
* Female partner with age 18-43 years
* Willing and able to give informed consent

Exclusion Criteria:

* Planned or performed diagnostic testicular biopsy (TESE) or percutaneous epididymal sperm aspiration (PESA)
* Use of donor-, cryopreserved- or electro-ejaculated semen
* Ovulation induction (OI) without IUI
* IVF for an absolute tubal factor
* Embryo-transfers after cryopreservation
* Embryo-transfer after pre-implantation genetic diagnosis
* Known genetic abnormalities related to infertility
* Known urological abnormality such as a varicocele or bilateral cryptorchism
* Use of other vitamin supplements

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1200 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 15 months
  Ongoing pregnancy ≥10-12 weeks of gestation

SECONDARY OUTCOMES:
Overall pregnancy rate | 15 months
  All pregnancies confirmed with a positive pregnancy (HCG) test
Time to pregnancy 1 - start intervention | 15 months
  The time between start of intervention and reaching ongoing pregnancy
Time to pregnancy 1 - start fertility treatment | 15 months
  The time between start of fertility treatment and reaching ongoing pregnancy
Change in semen parameters leading to change in treatment category | 15 months
  Between baseline and 3 months intervention, based on pre-wash total motile sperm count (TMSC) from the subpopulation from Radboudumc and sites that deliver a pre-wash TMSC before IUI/IVF/ICSI
Number of miscarriages | 15 months
  Defined as a non-vital intra-uterine pregnancy before 16 weeks of gestation
Live birth rate | 15 months
  Live birth rate defined as beyond 24 weeks of gestation, the birth of a living child.
Adverse effects | 15 months
  Gastro-intestinal problems such as reflux, obstipation, diarrhea, nausea or vomiting, furthermore loss of appetite, headache, dizziness, pruritus or skin rash.
Embryo fertilization rate | 15 months
  Relative improvement. Fertilization rate is the percentage of oocytes with >=2 PN after insemination (IVF) of injection (ICSI).
Embryo-utilization rate | 15 months
  Relative improvement of the embryo-utilization rate (EUR), defined as the number of high quality embryos obtained, embryo's used at transfer plus the number of embryos frozen, divided by the number of zygotes obtained in a cycle
Live birth rate | 15 months
  All live births

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek Nap, Prof.dr., Study Director — Gynecologist, head of department of Obstetrics and Gynaecology; Annemiek Nap, Prof MD PhD, Principal Investigator — Gynecologist, head of department of Obstetrics and Gynecology
Locations (21):
- Netherlands (21):
  - Fertiliteitscentrum Voorburg, Voorburg, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Maasziekenhuis Pantein, Boxmeer
  - Amphia ziekenhuis, Breda
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Nij Geertgen, Elsendorp
  - Treant ziekenhuis Scheper, Emmen
  - Nij Linge, Gorinchem
  - Medisch Centrum Kinderwens, Leiderdorp
  - Radboudumc, Nijmegen
  - Bravis Ziekenhuis, Roosendaal
  - Franciscus Gasthuis en Vlietland, Rotterdam
  - Maasstad ziekenhuis, Rotterdam
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Bernhoven Ziekenhuis, Uden
  - Máxima Medisch Centrum, Veldhoven
  - Nij Barrahus, Wolvega

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iwasaki A, Gagnon C. Formation of reactive oxygen species in spermatozoa of infertile patients. Fertil Steril. 1992 Feb;57(2):409-16. doi: 10.1016/s0015-0282(16)54855-9. PMID 1735495
- [Background] Zini A, de Lamirande E, Gagnon C. Reactive oxygen species in semen of infertile patients: levels of superoxide dismutase- and catalase-like activities in seminal plasma and spermatozoa. Int J Androl. 1993 Jun;16(3):183-8. doi: 10.1111/j.1365-2605.1993.tb01177.x. PMID 8359932
- [Background] Shekarriz M, Thomas AJ Jr, Agarwal A. Incidence and level of seminal reactive oxygen species in normal men. Urology. 1995 Jan;45(1):103-7. doi: 10.1016/s0090-4295(95)97088-6. PMID 7817460
- [Background] Agarwal A, Prabakaran S, Allamaneni S. What an andrologist/urologist should know about free radicals and why. Urology. 2006 Jan;67(1):2-8. doi: 10.1016/j.urology.2005.07.012. No abstract available. PMID 16413322
- [Background] Tremellen K. Oxidative stress and male infertility--a clinical perspective. Hum Reprod Update. 2008 May-Jun;14(3):243-58. doi: 10.1093/humupd/dmn004. Epub 2008 Feb 14. PMID 18281241
- [Background] Showell MG, Mackenzie-Proctor R, Brown J, Yazdani A, Stankiewicz MT, Hart RJ. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2014;(12):CD007411. doi: 10.1002/14651858.CD007411.pub3. Epub 2014 Dec 15. PMID 25504418
- [Background] Dattilo M, Cornet D, Amar E, Cohen M, Menezo Y. The importance of the one carbon cycle nutritional support in human male fertility: a preliminary clinical report. Reprod Biol Endocrinol. 2014 Jul 29;12:71. doi: 10.1186/1477-7827-12-71. PMID 25073983
- [Background] Dattilo M, D'Amato G, Caroppo E, Menezo Y. Improvement of gamete quality by stimulating and feeding the endogenous antioxidant system: mechanisms, clinical results, insights on gene-environment interactions and the role of diet. J Assist Reprod Genet. 2016 Dec;33(12):1633-1648. doi: 10.1007/s10815-016-0767-4. Epub 2016 Jul 16. PMID 27423667
- [Derived] de Ligny WR, de Bruin JP, Smits RM, Goovaerts IGF, Peeters K, Nap AW, Boxmeer JC, Donker RB, Schoonenberg M, Koks CAM, van Rumste MME, Visser J, Gielen SCJP, Boomsma CM, Smeenk JMJ, van Oppenraaij RHF, Cox T, Janse F, Muller LT, Brink-van der Vlugt JJ, Braat DDM, Fleischer K. Antioxidant Treatment and the Chance to Conceive in Men Seeking Fertility Care: The SUMMER Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2532405. doi: 10.1001/jamanetworkopen.2025.32405. PMID 40996763
- [Derived] Smits R, D'Hauwers K, IntHout J, Braat D, Fleischer K. Impact of a nutritional supplement (Impryl) on male fertility: study protocol of a multicentre, randomised, double-blind, placebo-controlled clinical trial (SUppleMent Male fERtility, SUMMER trial). BMJ Open. 2020 Jul 2;10(7):e035069. doi: 10.1136/bmjopen-2019-035069. PMID 32616489
- See also: Website Impryl — http://impryl.com/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03337360/Prot_SAP_001.pdf